CLINICAL TRIAL: NCT04759378
Title: Comorbid Disorders of the Esophagus in Patients With Irritable Bowel Disease
Brief Title: Comorbid Esophageal Disorders in IBS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bishoy Shehata, resident doctor at Assiut Univeristy Hospotal, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: esophageal disorders and IBS
Record Dates: First submitted 2021-01-12; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: GERD; Non-erosive Reflux Disease; Functional Esophageal Disorders; Irritable Bowel Syndrome
MeSH Terms: conditions — Gastroesophageal Reflux; Non-Erosive Reflux Disease; Irritable Bowel Syndrome | interventions — Gastroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBS patients who have upper GIT symptoms (Experimental)
  Interventions: Diagnostic Test: Upper endoscopy, esophageal manometry, 24-hour pH monitoring

INTERVENTIONS:
Diagnostic Test: Upper endoscopy, esophageal manometry, 24-hour pH monitoring — upper endoscopy determines if there are structural abnormalities in upper Git. esophageal manometry determines if there are motility disorders. 24-hour pH monitoring determines if acid reflux is present or not, and specifies its rate and duration.

SUMMARY:
assess the incidence of the entire spectrum of esophageal disorders and possible theories for overlap in IBS patients using different diagnostic modalities.

DETAILED DESCRIPTION:
In the practice of a gastroenterologist, irritable bowel syndrome (IBS) is the most frequent functional disorder. Its prevalence in the population is 9.8%-12.8%. Its frequency in women is more than men. In some studies, it has been shown that a patient may have an overlap of symptoms of different functional diseases of the gastrointestinal tract. Different researchers have ambiguously assessed the frequency of occurrence of esophageal disorders in patients with IBS. So, based on the publications of different authors, they are found in 15-80% of cases. In a study by N. de Bortoli et al. (2016) noted the association of IBS with functional heartburn in 77% of cases, and with GERD and hypersensitive esophagus (called heartburn associated with reflux) - in 33% of cases.

Traditionally, diagnostics of a combination of functional disorders of the esophagus and intestines were based on data X-ray and endoscopic methods. However modern research has shown the importance of using in this group of patients with daily combined pH impedance measurement. Thus, many authors have noted the undoubted advantages of this method in the diagnosis of esophageal disorders. Unfortunately, works devoted to this topic, extremely few in number, and the information obtained in them is quite contradictory, which indicates the need to continue research in this direction.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of IBS (according to the Rome criteria of the III revision).
* Upper GIT symptoms in the form of heartburn (sometimes belching), a lump in the throat, and non-cardiac chest pain.

Exclusion Criteria:

* History of thoracic, esophageal, or gastric surgery.
* Presence of duodenal or gastric ulcer on upper endoscopy.
* Presence of duodenal or gastric cancer on upper endoscopy.
* Conditions that prevent the installation of a nasogastric tube (nasopharyngeal formation, severe lumen-facial trauma).
* mental disorders state and disability.
* Pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-25 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of GERD in IBS patients who have upper GIT symptoms | baseline
  use the result of the comprehensive examination, upper endoscopy, esophageal manometry, and 24h pH monitoring to reveal that comorbid disorders of the esophagus in patients with IBS.
Incidence of Functional esophageal disorders in IBS patient who have upper GIT symptoms. | baseline
  use the result of the comprehensive examination, including upper endoscopy, esophageal manometry, and 24h pH monitoring to reveal that comorbid disorders of the esophagus in patients with IBS.